CLINICAL TRIAL: NCT01467492
Title: An Open-Label, Phase 4 Study of Telaprevir, Peginterferon Alfa-2a (Pegasys®), and Ribavirin (Copegus®) in Treatment-Experienced Black/African American and Non-Black/African American Subjects With Genotype 1 Chronic Hepatitis C Who Have Not Achieved a Sustained Viral Response With a Prior Course of Interferon-Based Therapy
Brief Title: Telaprevir, Peg-IFN-alfa-2a, and RBV in Treatment-Experienced Black/African American and Non-Black/African American Subjects With Genotype 1 Chronic Hepatitis C
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was decided by Sponsor on 13 January 2014 to terminate study early at primary efficacy endpoint as part of a decision to modify drug development plan.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-950-116
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C
Keywords: VX-950, Incivek
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black (Experimental): Telaprevir 750 milligram (mg) tablet 3 times per day for 12 weeks in combination with Peg-IFN-alfa-2a 180 microgram per week (mcg/week) subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 milligram per day (mg/day) (for participants weighing <75 kilograms [kg]) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Biological: Pegylated Interferon Alfa-2a
- Non-Black (Experimental): Telaprevir 750 mg tablet 3 times per day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day (for participants weighing <75 kg) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Biological: Pegylated Interferon Alfa-2a

INTERVENTIONS:
Drug: Telaprevir — Tablet
  Other Names: Incivek, VX-950
Drug: Ribavirin — Tablet
  Other Names: Copegus®, RBV
Biological: Pegylated Interferon Alfa-2a — Subcutaneous Injection
  Other Names: Pegasys®, Peg-IFN-Alfa-2a

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of telaprevir in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) and ribavirin (RBV) in treatment-experienced Black/African American and non-Black/African American participants with Genotype 1 Chronic Hepatitis C (CHC), who have not achieved a sustained viral response with a prior course of interferon-based therapy.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter study of treatment-experienced participants with Genotype 1 CHC, who self-identified as Black/African American (Group A) or who did not self-identify as Black/African American (Group B). Participants did not achieve a sustained virologic response 24 weeks after at least 1 prior course of Peg-IFN-alfa-2a/RBV therapy of standard duration, and have 1 of the following viral responses:

* Prior relapse: Participant had a documented undetectable hepatitis C virus ribonucleic acid (HCV RNA) level at the planned end of treatment of at least 42 weeks duration (HCV RNA evaluated anytime between 3 weeks before and 6 weeks after the last dose of Peg IFN-alfa-2a or RBV).
* Prior null response: Participant had a <2-log10 decrease in HCV RNA at 12 weeks, during prior Peg IFN-alfa-2a/RBV treatment, but never achieved undetectable HCV RNA while on treatment.
* Prior partial response: Participant had a >=2-log10 decrease in HCV RNA at 12 weeks, during prior Peg IFN-alfa-2a/RBV treatment, but never achieved undetectable HCV RNA while on treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants self-identify as Black/African American (Group A) or did not self-identify as Black/African American (Group B)
* Participants have Genotype 1 CHC and laboratory evidence of hepatitis C virus (HCV) infection for at least 6 months
* Participants did not achieve sustained viral response 24 weeks after last dose of study drug (SVR24), after at least 1 prior course of Peg-IFN-alfa-2a/RBV therapy of standard duration

Exclusion Criteria:

* Participants have received previous treatment with telaprevir or any other protease inhibitor(s) for CHC
* Participants who have evidence of hepatic decompensation
* Participants have diagnosed or suspected hepatocellular carcinoma
* Participants have any other cause of significant liver disease in addition to HCV
* Participants are currently abusing illicit drugs or alcohol, or have history of illicit substance or alcohol abuse within 2 years before the screening visit
* Participants who participated in any investigational drug study within 90 days before dosing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (27):
- United States (27):
  - Alabama, Birmingham, Alabama
  - California, San Francisco, California
  - Connecticut, New Haven, Connecticut
  - Washington, DC, Washington D.C., District of Columbia
  - Florida, Miami, Florida
  - Florida, Orlando, Florida
  - Florida, Tampa, Florida
  - Florida, West Palm Beach, Florida
  - Georgia, Atlanta, Georgia
  - Illinois, Chicago, Illinois
  - Louisiana, Baton Rouge, Louisiana
  - Louisiana, New Orleans, Louisiana
  - Louisiana, Shreveport, Louisiana
  - Maryland, Baltimore, Maryland
  - Massachusetts, Boston, Massachusetts
  - Michigan, Detroit, Michigan
  - New Jersey, Vineland, New Jersey
  - New York, New York, New York
  - New York, The Bronx, New York
  - North Carolina, Charlotte, North Carolina
  - North Carolina, Durham, North Carolina
  - Pennsylvania, Philadelphia, Pennsylvania
  - Texas, Dallas, Texas
  - Texas, Houston, Texas
  - Texas, San Antoinio, Texas
  - Virginia, Norfolk, Virginia
  - Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study included Prior Relapser (prior HCV treatment with pegylated interferon alfa/ribavirin [Peg-IFN/RBV] and experienced viral relapse) and Prior Null/Partial Responder (prior HCV treatment with Peg-IFN/RBV and had null/partial response) participants.
Pre-assignment Details: Efficacy analyses were reported as per Race (Black/Non-Black) (reporting arms) and also separately as per prior response (in categories) (Prior Relapser, Prior Null Responder, Prior Partial Responder as well as for Total Participants), unless otherwise specified.
Groups:
- Group A - Black: Black/African American participants received telaprevir 750 milligram (mg) tablet 3 times per day for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) (for participants weighing <75 kilograms [kg]) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
- Group B - Non-Black: Non-Black/African American participants received telaprevir 750 mg tablet 3 times per day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day (for participants weighing <75 kg) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
Period: Overall Study
Arm/Group | Group A - Black | Group B - Non-Black
Started | 83 | 38
Completed | 61 | 25
Not Completed | 22 | 13
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Study Terminated by Sponsor | 6 | 4
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Undefined | 2 | 0
Not completed — Enrolled But Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis (FA) Set included all enrolled participants who received at least 1 dose of any study drug.
Groups:
- Group A - Black: Black/African American participants received telaprevir 750 mg tablet 3 times per day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day (for participants weighing <75 kg) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Group A - Black | Group B - Non-Black | Total
Number analyzed (Participants) | 82 | 38 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (5.59) | 55.8 (5.95) | 57.1 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 6 | 40
  Male | 48 | 32 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response 12 Weeks After Last Actual Dose of Study Drug (SVR12)
Description: SVR12 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (<lower limit of quantification) at 12 weeks after last actual dose of study drug. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL).
Time Frame: 12 weeks after last actual dose of study drug (up to Week 60)
Population: FA Set. Here, n signifies participants who were evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  Prior Null Response (n = 41, 10) | 26.8 | 20.0
  Prior Partial Response (n= 20, 6) | 40.0 | 33.3
  Prior Relapse ( n= 21, 22) | 66.7 | 59.1
  Total (n= 82, 38) | 40.2 | 44.7

2. Secondary Outcome: Percentage of Participants With Sustained Viral Response 24 Weeks After Last Actual Dose of Study Drug (SVR24)
Description: SVR24 was defined as an undetectable HCV RNA Levels (<lower limit of quantification) at 24 weeks after last actual dose of study drug. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL.
Time Frame: 24 weeks after last actual dose of study drug (up to Week 72)
Population: FA Set. Here, n signifies participants who were evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  Prior Null Response (n = 41, 10) | 19.5 | 20.0
  Prior Partial Response (n= 20, 6) | 30.0 | 16.7
  Prior Relapse ( n= 21, 22) | 61.9 | 50.0
  Total (n= 82, 38) | 32.9 | 36.8

3. Secondary Outcome: Percentage of Participants With Extended Rapid Viral Response (eRVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. eRVR was defined as undetectable HCV RNA (<lower limit of quantification) at both 4 weeks and 12 weeks after the start of study treatment.
Time Frame: Week 4 and Week 12
Population: FA Set. Here, n signifies participants who were evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  Prior Null Response (n = 41, 10) | 24.4 | 30.0
  Prior Partial Response (n= 20, 6) | 45.0 | 66.7
  Prior Relapse ( n= 21, 22) | 66.7 | 68.2
  Total (n= 82, 38) | 40.2 | 57.9

4. Secondary Outcome: Percentage of Participants With Relapse
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. Relapse was defined as having undetectable HCV RNA (<lower limit of quantification) at actual end of treatment (EOT) and followed by detectable HCV RNA (>=lower limit of quantification) during follow-up.
Time Frame: 4 weeks (Wk) (up to Week 52), 12 weeks (up to Week 60) and 24 weeks (up to Week 72) after actual EOT
Population: FA Set. Here number of participants analyzed signifies participants with undetectable HCV RNA (HCV RNA <lower limit of quantification) at actual EOT and n signifies participants with undetectable HCV RNA at actual EOT for specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 48 | 26
percentage of participants
  Prior Null Response, 4 Wk After EOT (n=17,3) | 23.5 | 33.3
  Prior Null Response, 12 Wk After EOT (n=17,3) | 23.5 | 33.3
  Prior Null Response, 24 Wk After EOT (n=17,3) | 29.4 | 33.3
  Prior Partial Response, 4Wk After EOT (n=13,4) | 15.4 | 50.0
  Prior Partial Response, 12 Wk After EOT (n=13,4) | 23.1 | 50.0
  Prior Partial Response, 24 Wk After EOT (n=13,4) | 23.1 | 50.0
  Prior Relapse, 4 Wk After EOT (n=18,19) | 11.1 | 15.8
  Prior Relapse, 12 Wk After EOT (n=18,19) | 11.1 | 26.3
  Prior Relapse, 24 Wk After EOT (n=18,19) | 11.1 | 26.3
  Total, 4 Wk After EOT (n=48,26) | 16.7 | 23.1
  Total, 12 Wk After EOT (n=48,26) | 18.8 | 30.8
  Total, 24 Wk After EOT (n=48,26) | 20.8 | 30.8

5. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. Virologic breakthrough on treatment was defined as an increase of at least 1 log10 from nadir or confirmed detectable HCV RNA (>=lower limit of quantification) after undetectable HCV RNA (<lower limit of quantification). Percentages are calculated by using total number in FA set as denominator, in each category.
Time Frame: Week 2, 4, 8, and 12
Population: FA Set.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  Prior Null Response, Week 2 | 0 | 0
  Prior Null Response, Week 4 | 1.2 | 2.6
  Prior Null Response, Week 8 | 3.7 | 5.3
  Prior Null Response, Week 12 | 6.1 | 5.3
  Prior Partial Response, Week 2 | 0 | 0
  Prior Partial Response, Week 4 | 2.4 | 0
  Prior Partial Response, Week 8 | 2.4 | 0
  Prior Partial Response, Week 12 | 2.4 | 0
  Prior Relapse, Week 2 | 0 | 0
  Prior Relapse, Week 4 | 0 | 0
  Prior Relapse, Week 8 | 0 | 0
  Prior Relapse, Week 12 | 1.2 | 0
  Total, Week 2 | 0 | 0
  Total, Week 4 | 3.7 | 2.6
  Total, Week 8 | 3.7 | 5.3
  Total, Week 12 | 9.8 | 5.3

6. Secondary Outcome: Percentage of Participants With On Treatment Virologic Failure
Description: On treatment virologic failure was defined as meeting any futility rule or completing assigned treatment duration and having detectable HCV RNA at EOT. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. Futility rules: 1) Virologic breakthrough (at least 1 log10 increase from nadir or confirmed detectable HCV RNA after undetectable HCV RNA) from Day 1 through Week 24 or 48 (depending on treatment duration); 2) HCV RNA >1000 IU/mL during Weeks 4 to 12, inclusive; 3) Detectable HCV RNA after Week 12. Percentages are calculated by using total number in FA set as denominator, in each category.
Time Frame: Week 2, 4, 8, 12, 16, 24, 28, 36, 40, and 48
Population: FA Set.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  Prior Null Response, Week 2 | 0 | 0
  Prior Null Response, Week 4 | 4.9 | 2.6
  Prior Null Response, Week 8 | 8.5 | 7.9
  Prior Null Response, Week 12 | 12.2 | 7.9
  Prior Null Response, Week 16 | 19.5 | 7.9
  Prior Null Response, Week 24 | 23.2 | 10.5
  Prior Null Response, Week 28 | 23.2 | 13.2
  Prior Null Response, Week 36 | 25.6 | 13.2
  Prior Null Response, Week 40 | 28.0 | 13.2
  Prior Null Response, Week 48 | 29.3 | 13.2
  Prior Partial Response, Week 2 | 0 | 0
  Prior Partial Response, Week 4 | 2.4 | 0
  Prior Partial Response, Week 8 | 2.4 | 0
  Prior Partial Response, Week 12 | 4.9 | 0
  Prior Partial Response, Week 16 | 4.9 | 2.6
  Prior Partial Response, Week 24 | 6.1 | 7.9
  Prior Partial Response, Week 28 | 6.1 | 10.5
  Prior Partial Response, Week 36 | 7.3 | 10.5
  Prior Partial Response, Week 40 | 7.3 | 10.5
  Prior Partial Response, Week 48 | 7.3 | 10.5
  Prior Relapse, Week 2 | 0 | 0
  Prior Relapse, Week 4 | 0 | 0
  Prior Relapse, Week 8 | 0 | 0
  Prior Relapse, Week 12 | 1.2 | 0
  Prior Relapse, Week 16 | 1.2 | 0
  Prior Relapse, Week 24 | 1.2 | 2.6
  Prior Relapse, Week 28 | 1.2 | 2.6
  Prior Relapse, Week 36 | 1.2 | 2.6
  Prior Relapse, Week 40 | 1.2 | 5.3
  Prior Relapse, Week 48 | 1.2 | 5.3
  Total, Week 2 | 0 | 0
  Total, Week 4 | 7.3 | 2.6
  Total, Week 8 | 11.0 | 7.9
  Total, Week 12 | 18.3 | 7.9
  Total, Week 16 | 25.6 | 10.5
  Total, Week 24 | 30.5 | 21.1
  Total, Week 28 | 30.5 | 26.3
  Total, Week 36 | 34.1 | 26.3
  Total, Week 40 | 36.6 | 28.9
  Total, Week 48 | 37.8 | 28.9

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. AE includes SAE as well as Non-SAEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: Up to Week 52
Population: Safety Set.
Measure: Number; unit: percentage of participants
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 82 | 38
percentage of participants
  AE | 96.3 | 100.0
  SAE | 8.5 | 15.8

8. Secondary Outcome: Number of Participants With Telaprevir Resistant HCV Variant at Non-Structural Viral Protein 3-4A (NS3-4A) Region
Description: Sequence analysis of the HCV NS3-4A region was performed to monitor telaprevir-resistant variants. HCV RNA was isolated from the plasma, amplified by reverse transcription-polymerase chain reaction (RT-PCR), and sequenced (sequencing assay limit of detection HCV RNA >=1000 IU/mL). Results of this outcome measure were to be reported for overall participants instead of by race and by prior response.
Time Frame: up to Week 72
Population: FA Set.
Measure: Number; unit: participants
Groups:
- All Participants: All enrolled participants received telaprevir 750 mg tablet 3 times per day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day (for participants weighing <75 kg) or 1200 mg/day (for participants weighing >=75 kg) for 24 or 48 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 120
participants | 47

9. Other Pre Specified Outcome: Plasma Concentration of Telaprevir, Peginterferon Alfa-2a (Peg-IFN) and Ribavirin (RBV)
Time Frame: 48 weeks
Population: Pharmacokinetic sampling was not performed as per changes in planned analysis (protocol amendment); hence no data was collected.
Arm/Group | Group A - Black | Group B - Non-Black
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Arm/Group | Group A - Black | Group B - Non-Black
Serious Adverse Events (participants affected / at risk) | 7/82 | 6/38
Other Adverse Events (participants affected / at risk) | 79/82 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Black (N=82) | Group B - Non-Black (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Warm type haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Black (N=82) | Group B - Non-Black (N=38)
Fatigue (General disorders) | 31 | 26
Influenza like illness (General disorders) | 15 | 7
Injection site erythema (General disorders) | 9 | 4
Chills (General disorders) | 8 | 4
Pyrexia (General disorders) | 5 | 3
Injection site rash (General disorders) | 4 | 2
Asthenia (General disorders) | 2 | 3
Malaise (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 0 | 3
Chest pain (General disorders) | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Crying (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 0 | 1
Feeling jittery (General disorders) | 0 | 1
Injection site bruising (General disorders) | 0 | 1
Injection site discolouration (General disorders) | 1 | 0
Injection site discomfort (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 17
Anal pruritus (Gastrointestinal disorders) | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Haemorrhoids (Gastrointestinal disorders) | 8 | 5
Anorectal discomfort (Gastrointestinal disorders) | 8 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Vomiting (Gastrointestinal disorders) | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Haematochezia (Gastrointestinal disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 2
Cheilitis (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 2
Tongue discolouration (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oral lichen planus (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 16
Rash (Skin and subcutaneous tissue disorders) | 15 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 5 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 40 | 19
Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Headache (Nervous system disorders) | 14 | 13
Dizziness (Nervous system disorders) | 7 | 8
Dysgeusia (Nervous system disorders) | 4 | 3
Disturbance in attention (Nervous system disorders) | 2 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 3 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 10
Depression (Psychiatric disorders) | 8 | 4
Irritability (Psychiatric disorders) | 6 | 4
Anxiety (Psychiatric disorders) | 4 | 2
Sleep disorder (Psychiatric disorders) | 1 | 3
Mood swings (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Sinusitis (Infections and infestations) | 4 | 1
Cellulitis (Infections and infestations) | 3 | 1
Candida infection (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Carbuncle (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 3
Abnormal sensation in eye (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 1
Vitreous floaters (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Weight decreased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 1 | 1
Cardiac murmur (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 0
Amylase increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0
Penile discharge (Reproductive system and breast disorders) | 1 | 0
Penis disorder (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Flushing (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
It was decided by Sponsor on 13 January 2014 to terminate the study early as part of a decision to modify the drug development plan. Eligible participants completed virologic follow-up after termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.